CLINICAL TRIAL: NCT04311177
Title: Randomized Controlled Trial of Losartan for Patients With COVID-19 Not Requiring Hospitalization
Brief Title: Losartan for Patients With COVID-19 Not Requiring Hospitalization
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SURG-2020-28683
Record Dates: First submitted 2020-03-13; First posted 2020-03-17 (Actual); Results first posted 2022-05-04 (Actual); Last update posted 2022-05-04 (Actual); Status verified 2022-05

CONDITIONS: Corona Virus Infection; Acute Respiratory Distress Syndrome; SARS-CoV Infection
Keywords: COVID-19; Corona Virus; SARS-COV-2
MeSH Terms: conditions — Coronavirus Infections; Respiratory Distress Syndrome; Severe Acute Respiratory Syndrome; COVID-19 | interventions — Losartan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Losartan (Experimental): Participants in this arm will receive the study drug, Losartan.
  Interventions: Drug: Losartan
- Placebo (Placebo Comparator): Participants in this arm will receive a placebo treatment.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Losartan — Losartan; 25 mg daily; oral administration
  Other Names: Cozaar
  Arms: Losartan
Other: Placebo — Placebo (microcrystalline methylcellulose, gelatin capsule); oral administration
  Arms: Placebo

SUMMARY:
This is a multi-center, double-blinded study of COVID-19 infected patients randomized 1:1 to daily losartan or placebo for 10 days or treatment failure (hospital admission).

ELIGIBILITY:
Inclusion Criteria:

* Positive laboratory test for COVID-19 based on local laboratory standard
* Age greater than or equal to 18 years of age
* One of the following: Upper respiratory symptoms (cough, rhinorrhea) or fever (>101.5) or loss of taste / smell

Exclusion Criteria:

* Randomization > 72 hours of meeting inclusion criteria
* Randomization > 7 days of symptom onset
* Currently taking an angiotensin converting enzyme inhibitor (ACEi) or Angiotensin receptor blocker (ARB)
* Prior reaction or intolerance to an ARB or ACE inhibitor, including but not limited to angioedema
* Pregnant or breastfeeding women
* Females able to have children not currently taking a protocol allowed version of contraception: intrauterine device, Depo-formulation of hormonal contraception (e.g. medroxyprogesterone acetate/Depo-Provera), subcutaneous contraceptive (e.g. Nexplanon), daily oral contraceptives with verbalized commitment to taking daily throughout the study, condom use or abstinence during the study. All participants of child bearing potential enrolled in this fashion will be informed of the teratogenic risks.
* Patient reported history or electronic medical record history of kidney disease, defined as:

  1. Any history of dialysis
  2. History of chronic kidney disease stage IV
  3. Estimated Glomerular Filtration Rate (eGFR) of < 30ml/min/1.73 m2 (must be have been measured within 1 month of enrollment)
  4. Other kidney disease that in the opinion of the investigator, would affect losartan clearance
* Patient reported dehydration and significantly decreased urine output in the past 72 hours
* Most recent systolic blood pressure prior to enrollment <110 mmHg
* Patient reported history or electronic medical record history of severe liver disease, defined as:

  1. Cirrhosis
  2. History of hepatitis B or C
  3. Other liver disease that in the opinion of the investigator, would affect losartan clearance
  4. Documented AST or ALT > 3 times the upper limit of normal within 3 months of randomization (if available in electronic medical record)
* Potassium >5.0 mmol/L (must have been measured within 1 month) of enrollment
* Concurrent treatment with aliskiren
* Inability to obtain informed consent
* Enrollment in another blinded randomized clinical trial for COVID

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 117 (Actual)
Dates: Start 2020-04-09 (Actual); Primary Completion 2021-02-01 (Actual); Study Completion 2021-02-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Tignanelli, MD, Principal Investigator — University of Minnesota; Michael Puskarich, MD, MS, Principal Investigator — University of Minnesota
Locations (4):
- United States (4):
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - M Health Fairview University of Minnesota Medical Center, Minneapolis, Minnesota
  - University of Minnesota, Minneapolis, Minnesota
  - Mayo Clinic Health System, Rochester, Minnesota

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Puskarich MA, Cummins NW, Ingraham NE, Wacker DA, Reilkoff RA, Driver BE, Biros MH, Bellolio F, Chipman JG, Nelson AC, Beckman K, Langlois R, Bold T, Aliota MT, Schacker TW, Voelker HT, Murray TA, Koopmeiners JS, Tignanelli CJ. A multi-center phase II randomized clinical trial of losartan on symptomatic outpatients with COVID-19. EClinicalMedicine. 2021 Jun 17;37:100957. doi: 10.1016/j.eclinm.2021.100957. eCollection 2021 Jul. PMID 34195577
- [Derived] Smolander J, Bruchfeld A. [COVID-19 and kidney disease]. Lakartidningen. 2020 Jul 13;117:20110. Swedish. PMID 32658300

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Losartan | Placebo
Started | 58 | 59
Completed | 50 | 55
Not Completed | 8 | 4
Not completed — Adverse Event | 3 | 1
Not completed — Physician Decision | 4 | 3
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Losartan | Placebo | Total
Number analyzed (Participants) | 58 | 59 | 117
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 55 | 59 | 114
  >=65 years | 3 | 0 | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33 | 25 | 58
  Male | 25 | 34 | 59
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 5 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 4 | 8
  White | 45 | 40 | 85
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 8 | 10 | 18

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Admitted to the Hospital
Description: Outcome reported as the percentage of participants per arm admitted to inpatient hospital care due to COVID-19-related disease within 15 days of randomization.
  Currently, there is a pre-planned pooled analysis with a national trial network under development.
Time Frame: 15 days
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Losartan | Placebo
Number analyzed (Participants) | 58 | 59
percentage of participants | 5.2 [1.1 to 14.4] | 1.7 [0.0 to 9.1]

2. Secondary Outcome: Change in PROMIS Dyspnea Scale
Description: The PROMIS dyspnea scale consists of 4 subscales. 3 (1. general shortness of breath, 2. intensity, and 3. Frequency) are scored from 0 (no symptoms) to 10 (most severe). The 4th subscale is scored from 0-4 in response to the question "I've been short of breath" with 0 representing none and 4 the most severe, for a total range of 0-34. Results are difference between enrollment and day 10. There are no units.
Time Frame: 10 days
Population: Only 50 patients were analyzed for this outcome measure due to loss to follow-up or refusal to complete the survey resulting in data missingness.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Losartan | Placebo
Number analyzed (Participants) | 50 | 50
score on a scale | -0.4 (0.9) | -0.5 (0.7)

3. Secondary Outcome: Change in SF-12 Physical Composite Score
Description: The SF-12 is a self-reported validated outcome measure assessing the impact of health on an individual's everyday life. Patients fill out a 12 question survey which is then scored by a clinician or researcher. Physical score is computed using the scores of twelve questions and range from 0 to 100, where a zero score indicates the lowest level of health measured by the scales and 100 indicates the highest level of health. The 33-item Severity bank assesses the severity of difficulty breathing during various specific activities (the same 33 activities assessed in Dyspnea Functional Limitations). Each activity is rated in terms of degree of dyspnea (0 = no shortness of breath, 1 = mildly short of breath, 2 = moderately short of breath, 3 = severely short of breath) while engaging in the activity over the past 7 days. Total scores range from 0 to 99 with higher scores reflecting greater levels of dyspnea during daily activity.
Time Frame: 10 days
Measure: Mean (Standard Deviation); unit: score
Arm/Group | Losartan | Placebo
Number analyzed (Participants) | 31 | 39
score | 1.4 (9.1) | 0.2 (6.5)

4. Secondary Outcome: Change in SF-12 Mental Composite Score
Description: The SF-12 is a self-reported validated outcome measure assessing the impact of health on an individual's everyday life. Patients fill out a 12 question survey which is then scored by a clinician or researcher. Mental composite score is computed using the scores of twelve questions and range from 0 to 100, where a zero score indicates the lowest level of health measured by the scales and 100 indicates the highest level of health.
Time Frame: 10 days
Measure: Mean (Standard Deviation); unit: score
Arm/Group | Losartan | Placebo
Number analyzed (Participants) | 31 | 39
score | -0.1 (6.5) | -0.3 (5.7)

5. Secondary Outcome: Daily Maximum Temperature
Description: Participants will report their maximum daily oral temperature to the study team. Outcome is reported as the mean maximum daily body temperature (in degrees Celsius) over 10 days.
Time Frame: 10 days
Measure: Mean (Standard Error); unit: degrees Farenheit
Arm/Group | Losartan | Placebo
Number analyzed (Participants) | 58 | 59
degrees Farenheit | 97.7 (0.097) | 97.8 (0.092)

6. Secondary Outcome: Count of Participants With an Emergency Department or Clinic Presentation
Description: Outcome is reported as the mean number of emergency department and clinic presentations combined per participant in each arm.
Time Frame: 28 days
Measure: Count of Participants; unit: Participants
Arm/Group | Losartan | Placebo
Number analyzed (Participants) | 58 | 59
Participants | 10 | 5

7. Secondary Outcome: Disease Severity Rating Day 15
Description: Outcome reported as the number of participants in each arm who fall into each of 7 categories. Lower scores indicate greater condition severity. The ordinal scale is an assessment of the clinical status at the first assessment of a given study day. The scale is as follows: 1) Death; 2) Hospitalized, on invasive mechanical ventilation or extracorporeal membrane oxygenation (ECMO); 3) Hospitalized, on non-invasive ventilation or high flow oxygen devices; 4) Hospitalized, requiring supplemental oxygen; 5) Hospitalized, not requiring supplemental oxygen; 6) Not hospitalized, limitation on activities; 7) Not hospitalized, no limitations on activities.
Time Frame: 15 days
Measure: Mean (Standard Deviation); unit: score
Arm/Group | Losartan | Placebo
Number analyzed (Participants) | 58 | 59
score | 5.8 (0.5) | 5.9 (0.7)

8. Secondary Outcome: Change in Viral Load by Nasopharyngeal Swab at Day 9
Description: Viral load is measured as number of viral genetic copies per mL.
Time Frame: 9 days
Measure: Mean (Standard Error); unit: log10 copies/mL
Arm/Group | Losartan | Placebo
Number analyzed (Participants) | 32 | 35
log10 copies/mL | -3.8 (0.3) | -3.6 (0.29)

9. Secondary Outcome: Change in Viral Load by Nasopharyngeal Swab at Day 15
Description: Viral load is measured as number of viral genetic copies per mL.
Time Frame: 15 days
Measure: Mean (Standard Error); unit: log10 copies/mL
Arm/Group | Losartan | Placebo
Number analyzed (Participants) | 35 | 25
log10 copies/mL | -3.7 (0.33) | -4 (0.29)

10. Secondary Outcome: Percentage of Patients Admitted to the Intensive Care Unit Within 15 Days
Description: Outcome reported as the percent of participants in each arm who require ICU admission by day 15 following randomization.
Time Frame: 15 days
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Losartan | Placebo
Number analyzed (Participants) | 58 | 59
percentage of participants | 1.7 [0.0 to 9.2] | 1.7 [0.0 to 9.1]

11. Secondary Outcome: Need for Oxygen Therapy at 15 Days
Description: Outcome reported as the percent of participants in each arm who require oxygen therapy by day 15 following randomization.
Time Frame: 15 days
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Losartan | Placebo
Number analyzed (Participants) | 58 | 59
percentage of participants | 1.7 [0.0 to 9.2] | 1.7 [0.0 to 9.1]

ADVERSE EVENTS:
Time Frame: 28 days
Description: Events were monitored / assessed without regard to specific adverse event term, but rather by systems.
Arm/Group | Losartan | Placebo
All-Cause Mortality (participants affected / at risk) | 0/58 | 0/59
Serious Adverse Events (participants affected / at risk) | 3/58 | 1/59
Other Adverse Events (participants affected / at risk) | 43/58 | 56/59
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Losartan (N=58) | Placebo (N=59)
Hospital Admission (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Losartan (N=58) | Placebo (N=59)
Cardiovascular (Cardiac disorders) | 9 (9) | 6 (6)
Constitutional (Social circumstances) | 6 (6) | 13 (13)
Ear, Nose, and Throat (Ear and labyrinth disorders) | 7 (7) | 4 (4)
Gastrointestinal (Gastrointestinal disorders) | 4 (4) | 4 (4)
Neurologic (Nervous system disorders) | 3 (3) | 2 (2)
Renal (Renal and urinary disorders) | 2 (2) | 5 (5)
Respiratory (Respiratory, thoracic and mediastinal disorders) | 9 (9) | 22 (22)
Skin (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-04-05): https://cdn.clinicaltrials.gov/large-docs/77/NCT04311177/Prot_SAP_000.pdf
  • Informed Consent Form (2020-04-07): https://cdn.clinicaltrials.gov/large-docs/77/NCT04311177/ICF_002.pdf